CLINICAL TRIAL: NCT04824118
Title: Measuring the Changes in Clotting Parameters Before and After Medical Abortion
Brief Title: Clotting Parameters After Medical Abortion
Acronym: C-PLAN
Status: Completed | Type: Observational
Sponsor: NHS Lothian (Other Government)
Collaborators: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC20164
Record Dates: First submitted 2020-12-07; First posted 2021-04-01 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Abortion Early; Abortion, Complete; Abortion, Second Trimester; Termination of Pregnancy Complicated by Embolism; Venous Thromboses; Venous Thromboembolism; Venous Thromboembolic Disease; Clotting Disorder
MeSH Terms: conditions — Venous Thrombosis; Venous Thromboembolism; Hemostatic Disorders | interventions — Thrombelastography; Blood Cell Count; Pregnancy Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples - testing for clotting factors
  Urine - point of care pregnancy test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Gestation less than 10 weeks: Blood tests and urine sample at baseline and 10-14 days after mifepristone administration
  Interventions: Diagnostic Test: Thromboelastometry; Diagnostic Test: Clotting Studies; Diagnostic Test: Full Blood Count; Diagnostic Test: Quantitative hCG
- Group 2: Gestation 10-14 weeks: Blood tests and urine sample at baseline and 10-14 days after mifepristone administration
  Interventions: Diagnostic Test: Thromboelastometry; Diagnostic Test: Clotting Studies; Diagnostic Test: Full Blood Count; Diagnostic Test: Quantitative hCG
- Group 3: Gestation 14-20 weeks: Blood tests and urine sample at baseline and 10-14 days after mifepristone administration
  Interventions: Diagnostic Test: Thromboelastometry; Diagnostic Test: Clotting Studies; Diagnostic Test: Full Blood Count; Diagnostic Test: Quantitative hCG
- Group 4: Non-pregnant controls: Blood tests at baseline only.
  Interventions: Diagnostic Test: Thromboelastometry; Diagnostic Test: Clotting Studies; Diagnostic Test: Full Blood Count; Diagnostic Test: Pregnancy Test

INTERVENTIONS:
Diagnostic Test: Thromboelastometry — Point of Care Test for clotting parameters (ClotPro device)
Diagnostic Test: Clotting Studies — Standard laboratory tests for clotting:
  * International normalised ratio (INR)
  * Prothrombin time (PT)
  * adjusted partial thromboplastin time (aPTT)
  * fibrinogen
Diagnostic Test: Full Blood Count — For platelet count
Diagnostic Test: Quantitative hCG — Serum human chorionic gonadotrophin
  Groups: Group 1: Gestation less than 10 weeks; Group 2: Gestation 10-14 weeks; Group 3: Gestation 14-20 weeks
Diagnostic Test: Pregnancy Test — Point of care urinary pregnancy test
  Groups: Group 4: Non-pregnant controls

SUMMARY:
Venous thromboembolism (VTE - blood clots that form in deep veins or in the lungs) has been identified as a leading cause of death in economically developed countries for pregnant and recently-pregnant women.

There is evidence that clotting parameters can take up to 6 weeks to return to normal for women who have had term deliveries, however there is an absence of information on time taken for clotting parameters to normalise following abortion.

As such, existing guidelines are based solely on expert opinion and recommend durations of VTE prevention from as short as 7 days, up to 6 weeks following abortion.

All women are assessed for risk of VTE, but data are needed to inform an evidence-based approach to prevention of VTE in these women.

The findings from this pilot study have the potential to inform clinical guidance and possibly a larger study subsequently.

DETAILED DESCRIPTION:
Sample population: Women who attend the abortion service at the Chalmers Centre to receive abortion assessment and abortion care. There will be 3 groups recruited based upon gestational age of pregnancy - Group 1: Gestation less than 10 weeks (10 participants), Group 2: Gestation 10+0 -13+6 weeks (10 participants), Group 3: Gestation 14+0-20+0 weeks (10 participants).

Information Sheet: All new patients attending the clinic will be given a copy of the participant information sheet, so that they have time to read about the study. The Information sheet will also be available on the 'research' section of the clinic website - all women are routinely directed to this page before attending clinic.

Approach by research staff: Following registration, all patients are taken for an ultrasound scan by a clinical support worker to confirm gestation. Following this, patients move to a waiting area until they can be seen for their assessment. While they are waiting, the clinic coordinator will ask the patient if they are happy to be approached by the researcher to discuss the study further. If they are happy to discuss further, the researcher will then approach and discuss the study in a private room.

Consent: If patients are happy to participate in the study, the researcher will then obtain written informed consent prior to their bloods being taken by clinic staff if bloods required for routine care, if no routine bloods are required, the researcher will obtain the blood sample. Participants will be asked if they are planning to use a hormonal form of contraception following their abortion - if yes, they would be asked to wait until they have had their second blood sample taken to commence or not taken forward into the study.

First blood test: This will be obtained on the day of clinic attendance and ultrasound scan. Blood samples (less than 20 ml) will be obtained and taken to the NHS Lothian laboratory at the Royal Infirmary of Edinburgh and for ClotPro thromboelastography point of care testing.

Second blood test: An appointment will be made to see the patient in Chalmers Centre or at their home to obtain a further blood sample to compare to the initial test. This will take place 10-14 days following mifepristone administration. For the repeat sample we will conduct a COVID-19 risk assessment and only invite them for return visit/home visit if:

1. The participant has confirmed they and close contacts are well and without suspicion of COVID-19.
2. The participant agrees to a home visit.
3. The research staff undertaking the home visit should be well and have had no known contact with a COVID-19 positive individual for the past 14 days.

If they are having an intrauterine contraceptive, implant or injection, the second blood sample can be taken when they come into clinic for this, to minimise the number of visits.

Comparison group: A comparison group, Group 4 (10 participants), who are healthy volunteers, recruited from sexual and reproductive health clinics at Chalmers Centre, will be asked to provide a single blood test for ClotPro and lab tests, and urine pregnancy test hCG to act as a nonpregnant comparison. These participants must not be using hormonal contraception and must not be pregnant. This group will be approached by clinicians working in the SRH clinics and the researcher will be on hand to obtain consent and then draw blood.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* Pregnant and seeking abortion
* Gestation of pregnancy less than 10 weeks
* Healthy, no medical conditions

Group 2:

* Pregnant and seeking abortion
* Gestation of pregnancy between 10 and 14 weeks
* Healthy, no medical conditions

Group 3:

* Pregnant and seeking abortion
* Gestation of pregnancy between 14 to 20 weeks
* Healthy, no medical conditions

Group 4:

* Non pregnant
* Healthy, no medical conditions
* Able to speak English independently

Exclusion Criteria:

All groups:

* Unable to give informed consent
* Previous or current venous thromboembolism
* Current smoker
* Personal or family history of thrombophilia or haemophilia
* Taking medicines known to affect clotting parameters (e.g. Aspirin)

Groups 1-3:

- Planning to commence hormonal contraception prior to second blood test.

Group 4:

- Using hormonal contraception at baseline visit

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Cisgendered women. Non-binary assigned female at birth and transgendered men would be considered as long as they are not using any hormonal therapy (cross-sex, blockers or otherwise)
Study Population: Women seeking medical abortion at various gestations and non-pregnant comparator group.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
Clotting Time in Seconds | 10-14 days
  As measured using ClotPro device between baseline and follow up for Groups 1-3.
Clot Formation Time in Seconds | 10-14 days
  As measured using ClotPro device between baseline and follow up for Groups 1-3.
Maximal Amplitude in millimeters | 10-14 days
  On clotting curve as measured using ClotPro device between baseline and follow up for Groups 1-3.
Maximum Lysis of clot in percentage | 10-14 days
  As measured using ClotPro device between baseline and follow up for Groups 1-3.
Clot Lysis index in percentage | 10-14 days
  As measured using ClotPro device between baseline and follow up for Groups 1-3.
Lysis time in seconds | 10-14 days
  As measured using ClotPro device between baseline and follow up for Groups 1-3.

SECONDARY OUTCOMES:
Prothrombin Time in seconds | 10-14 days
  Assessed by laboratory tests between baseline and follow up in Groups 1-3 and in comparison with group 4.
Activated Partial Thromboplastin Time in seconds | 10-14 days
  Assessed by laboratory tests between baseline and follow up in Groups 1-3 and in comparison with group 4.
International Normalised Ratio (INR) | 10-14 days
  Assessed by laboratory tests between baseline and follow up in Groups 1-3 and in comparison with group 4.
Fibrinogen in grams per litre | 10-14 days
  Assessed by laboratory tests between baseline and follow up in Groups 1-3 and in comparison with group 4.
Platelet count (x10^9 per litre) | 10-14 days
  Assessed by laboratory tests between baseline and follow up in Groups 1-3 and in comparison with group 4.
Thromboelastography parameters (comparison with non-pregnant group) | 10-14 days
  Comparison of thromboelastography parameters (as measured using ClotPro device) between Groups 1-3 with Group 4.
Serum hCG in units per litre | 10-14 days
  Comparison of serum hCG levels between baseline and follow up in groups 1-3
Lysis time in seconds | 10-14 days
  As measured using ClotPro device between baseline and follow up for Groups 1-3.
Clot Lysis index in percentage | 10-14 days
  As measured using ClotPro device comparing Groups 1-3 with Group 4
Maximum Lysis of clot in percentage | 10-14 days
  As measured using ClotPro device comparing Groups 1-3 with Group 4
Maximal Amplitude in millimeters | 10-14 days
  As measured using ClotPro device comparing Groups 1-3 with Group 4.
Clot Formation Time in Seconds | 10-14 days
  As measured using ClotPro device comparing Groups 1-3 with Group 4
Clotting Time in Seconds | 10-14 days
  As measured using ClotPro device comparing Groups 1-3 with Group 4

CONTACTS AND LOCATIONS:
Overall Officials: John J Reynolds-Wright, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- Chalmers Centre for Sexual and Reproductive Health, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
As this is abortion-care research with small numbers of participants, we will not make individual level participant data available publicly. Should researchers required this data for meta-analysis (for example) they can contact the principle investigator and request will be considered on a case-by-case basis.